CLINICAL TRIAL: NCT01884662
Title: Virtual Walking for Reducing Spinal Cord Injury-Related Neuropathic Pain
Brief Title: Virtual Walking for Neuropathic Pain in Spinal Cord Injury
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, John S. Richards, Principal Investigator, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: H133N110008VWalking
Record Dates: First submitted 2012-09-11; First posted 2013-06-24 (Estimated); Last update posted 2021-08-30 (Actual); Status verified 2021-08

CONDITIONS: Spinal Cord Injury; Neuropathic Pain
Keywords: spinal cord injury; neuropathic pain
MeSH Terms: conditions — Spinal Cord Injuries; Neuralgia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Virtual walking (Experimental): A 3D video of legs walking from a first person perspective have been developed in consultation with persons with SCI and virtual reality experts. Participants are provided with a 3D monitor and Blue Ray player for daily viewing of the tape for two weeks.
  Interventions: Behavioral: Virtual walking
- Wheeling tape (Active Comparator): A 3D video was produced of legs in a wheelchair covering the identical conditions of the walking experimental video.
  Interventions: Behavioral: Wheeling tape

INTERVENTIONS:
Behavioral: Virtual walking — As in mirror therapy for amputee phantom pain, there is evidence that neuropathic SCI pain responds to images of the person with SCI's legs "walking"; we achieve this via a virtual reality approach where the subject perceives it is his/her legs walking.
  Arms: Virtual walking
Behavioral: Wheeling tape — This control condition mirrors the experimental condition in all respects except it shows still legs in a wheelchair traversing the same path as the virtual walking condition
  Other Names: A video of a person's legs in a wheelchair traversing a path
  Arms: Wheeling tape

SUMMARY:
Spinal cord injury neuropathic pain (SCI-NP) is a common problem, and when severe, is one of the most problematic of secondary conditions that is minimally to modestly responsive to currently available treatments. It is usually described as burning or stabbing, and is located at or below the level at which their sensation changes from normal to impaired; persons with no feeling at all in their legs for example can experience pain in the legs. The purpose of this project is to further investigate the use of a novel visual stimulation treatment; a technique that has shown benefit in other populations with chronic pain secondary to deafferentation. To accomplish this, a novel treatment - virtual reality (VR) walking - will be examined. Should this treatment show benefit, a portable, accessible means of treatment will be available for persons with SCI and for whom transportation to health care providers is often difficult.

DETAILED DESCRIPTION:
This treatment will be investigated in two-phase project:

Phase 1: Determine the efficacy of VR treatments as a home-based approach and determine the effect of VR treatment on reversal of maladaptive cortical reorganization associated with SCI-NP, as has been shown in other populations with neuropathic pain secondary to deafferentation.

Phase 2: Determine the effectiveness and immediate analgesic effect of VR treatment among persons with both tetraplegia and paraplegia.

The primary outcome variable of this research is the severity of SCI-NP with a secondary outcome of level of pain interference with daily activities.

In the phantom pain literature for persons with amputations, treatment paradigms based on visual stimulation, called mirror therapies, have proven helpful. These approaches involve the person viewing a mirror image of their intact limb to produce the visual illusion of a return of the missing limb, often with a marked reduction in pain following. Investigations have demonstrated that such approaches reduce pain in some individuals and that this change is associated with reversal of the functional reorganization in the somatosensory cortex. There has been one study of neuropathic pain in SCI that demonstrated good neuropathic pain relief with a mirror image of the upper half of the individual with SCI with the lower half of their body represented by a rear projection screen generated image of walking legs. We have collaborated with this author, and developed and pilot tested a virtual walking DVD that is presented via virtual reality goggles to enhance the first person sense of immersion. Results were sufficiently encouraging to cause us to seek funding for current, broader project

ELIGIBILITY:
Inclusion Criteria: traumatic onset SCI, at least three months post onset, between 19 and 65; at least 6th grade reading level; neuropathic pain averaging at least 4/10.

-

Exclusion Criteria: Unable to independently transfer to the fMRI scanning table, current pressures sores, contraindications to scanning; non-compliance with a pre-assignment task.

-

Ages: 19 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2012-09 (Actual); Primary Completion 2021-04-30 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
Changes in Numeric Rating Scale | Baseline, post 14 day treatment, one week, one month, three months, 6 months post 14 day treatment. Changes in the NRS scale will be the outcome
  The NRS is the most commonly used pain rating scale, and ranges from 0/10 to 10/10 with 10 representing unbearable or the "worst possible pain".

SECONDARY OUTCOMES:
Changes in fMRI correlates of neuropathic pain | Baseline and immediately post 14 day treatment
  We will use CASL-fMRI image processing and methods for estimating shifts in cortical somatosensory plasticity
Changes in Pain Interference | Baseline, immediately post 14 day treatment, one week, and one, three and six months post treatment
  The seven pain interference items of the Brief Pain Inventory
Changes in Neuropathic Pain Scale | Baseline, immediately 14 days post treatment, one week, one, three and six months post treatment
  An 11 item scale specifically measuring the symptoms of neuropathic pain.

CONTACTS AND LOCATIONS:
Overall Officials: John S Richards, PhD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- Spain REhabilitation Center, Birmingham, Alabama, United States

REFERENCES:
- [Derived] Richardson EJ, McKinley EC, Rahman AKMF, Klebine P, Redden DT, Richards JS. Effects of virtual walking on spinal cord injury-related neuropathic pain: A randomized, controlled trial. Rehabil Psychol. 2019 Feb;64(1):13-24. doi: 10.1037/rep0000246. Epub 2018 Nov 8. PMID 30407030